CLINICAL TRIAL: NCT05085132
Title: An Efficacy Trial of the MindFi App for Stress, Well-being, and Sleep Quality in Working Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Jaedye Labs (Unknown)
Responsible Party: Principal Investigator, Julian Lim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MINDFI01
Record Dates: First submitted 2021-09-22; First posted 2021-10-20 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Stress; Burnout
Keywords: Mindfulness; Sleep quality; Well-being
MeSH Terms: conditions — Burnout, Psychological; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 allocation to use the MindFi app or receive a dummy version of the app (containing music tracks for relaxation).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MindFi app: Standard content (Experimental): Participants will receive full access to the MindFi app, containing learning tracks, practice tracks, and assessments. Participants will be instructed to use a practice track for a minimum of 10 minutes a day, and may use other exercises or tracks if desired. The intervention will last 4 weeks.
  Interventions: Behavioral: MindFi app: Standard content
- Mindfi app: Standard content without practice (Sham Comparator): Participants will receive full access to the MindFi app, containing learning tracks, music tracks, and assessments. Participants will be instructed to use a music track for a minimum of 10 minutes a day, and may use other exercises or tracks if desired. The intervention will last 4 weeks.
  Interventions: Behavioral: Mindfi app: Standard content without practice

INTERVENTIONS:
Behavioral: MindFi app: Standard content — Digital wellness training in this study will be delivered via the MindFi app, designed by Jaedye Labs. Content includes learning, assesesment, and practice tracks A core component of the exercises in this app is mindfulness training; however, the app also incorporates other exercises drawn from positive psychology such as journaling and diaphragmatic breathing. The app goes beyond traditional guided meditation through content that reinforces the principles and attitudes taught during in-person training, and also seeks to maximize user experience by using interactive tasks and progress charts.
  Arms: MindFi app: Standard content
Behavioral: Mindfi app: Standard content without practice — In this condition, participants will receive a version of the MindFi app that does NOT contain the practice tracks, only the learning and assessment tracks.
  Arms: Mindfi app: Standard content without practice

SUMMARY:
90% of Asian workers report high levels of stress in an "always-on" culture. Stress and burnout are risk factors that account for 10-20% of health expenditure and threaten work longevity in the world's fastest growing economies. Traditional face-to-face sources of mental care such as counseling and psychotherapy are effective as a countermeasure to stress, but not always accessible or acceptable for those with busy lifestyles. Because of this, there is an urgent need for on-demand, scalable interventions to reduce stress and improve mental and physical well being. Technology-based solutions are increasingly being proposed to fill this need.

MindFi is a smartphone app that uses mindfulness exercises to help users cope with work stress and increase productivity. Since 2017, it has been featured by Apple, BBC, and Bloomberg and is being used at corporates such as Bain, Bloomberg, Cigna, and Zendesk. MindFi users contribute behavioral and self-report data, which are then used to generate individual recommendations for relevant, evidence-based exercises. These include mental care techniques such as mindfulness meditation, therapeutic journaling, psychosocial support and educational wellbeing quizzes.

In this study, the investigators will recruit 200 participants in a randomized controlled design, with 100 receiving access to content of the MindFi app, and 100 receiving access to a version containing music tracks for relaxation. Each intervention will last 4 weeks. Participants will use these apps for a period of 5 weeks (for a minimum of 10 minutes per day). Pre- and post-intervention, the investigators will measure self-reported ratings on a number of psychological variables, and will track sleep quality objectively for a one-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Currently in full-time employment
2. Fluent in English
3. DASS-21 scores of at least 10 on the Stress subscale

Exclusion Criteria:

1. Current diagnosis of a chronic psychological disorder, or sleep disorder
2. Regularly practising meditation

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
WHO Well-Being Index (WHO, 1998) | Week 0 (at the start of the intervention) and Week 5
  Change in self-reported mental well being (min score: 0; max score: 25; greater increases in this score represent a better outcome)
Depression, Anxiety, And Stress Scale -- Stress subscale (Lovibond and Lovibond, 1985) | Week 0 (at the start of the intervention) and Week 5
  Change in self-report measure of stress (min score: 0; max score: 21; greater reductions in this score represent a better outcome)
Change in Sleep Efficiency (Oura Ring) | Week 0 (at the start of the intervention) and Week 5
  (Latency + wake time)/Time in bed, as calculated by the Oura app

SECONDARY OUTCOMES:
Depression, Anxiety, And Stress Scale -- Depression subscale (Lovibond and Lvibond, 1985) | Week 0 (at the start of the intervention) and Week 5
  Change in Self-report measure of depression (min score: 0; max score: 21; greater reductions in this score represent a better outcome)
Depression, Anxiety, And Stress Scale -- Anxiety subscale (Lovibond and Lvibond, 1985) | Week 0 (at the start of the intervention) and Week 5
  Change in Self-report measure of anxiety (min score: 0; max score: 21; greater reductions in this score represent a better outcome)
Maslach Burnout Inventory (Maslach et al., 1996) | Week 0 (at the start of the intervention) and Week 5
  Change in self-report measure of burnout
  3 subscales:
  1. Emotional exhaustion (min score: 0; max score: 54; greater reductions in this score represent a better outcome)
  2. Depersonalization (min score: 0; max score: 30; greater reductions in this score represent a better outcome)
  3. Personal achievement (min score: 0; max score: 48; greater increases in this score represent a better outcome)
Five Factor Mindfulness Questionnaire (Baer et al., 2006) | Week 0 (at the start of the intervention) and Week 5
  Change in Self-report measure of trait mindfulness (min score: 39; max score: 195; greater increases in this score represent a better outcome)
Brief Inventory of Thriving (Su et al., 2014) | Week 0 (at the start of the intervention) and Week 5
  Change in Self-report measure of eudaimonic well-being (min score: 10; max score: 50; greater increases in this score represent a better outcome)
Resting heart rate during sleep (from Oura Ring) | Week 0 (at the start of the intervention) and Week 5
  Objective measure of resting heart rate
Heart-rate variability during sleep (from Oura Ring) | Week 0 (at the start of the intervention) and Week 5
  Objective measure of heart rate variability
Satisfaction with Life Scale (Diener et al., 1985) | Week 0 (at the start of the intervention) and Week 5
  Self-report measure of hedonic well being (min score: 5; max score: 35; greater increases in this score represent a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Lim, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared with other researchers upon reasonable request, and after publication of the study results,
Supporting Information: ICF, Analytic Code
Time Frame: The data will become available after publication into perpetuity.
Access Criteria: Researchers with a reasonable re-analysis plan will be eligible for data sharing